CLINICAL TRIAL: NCT05196607
Title: Degrees of New Information and Communication Technologies (ICT) Use Among Surgical Patients (NINASPA Study)
Brief Title: Degrees of New ICT Use Among Surgical Patients
Acronym: NINASPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Jose-M Ramirez, Prof, Universidad de Zaragoza
Other Study IDs: UZaragoza-2
Record Dates: First submitted 2021-12-29; First posted 2022-01-19 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Surgery, Elderly patient, New technologies
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A dedicated survey on the use of mobile applications to all patients who were to be operated on a scheduled basis in our Surgery Service

SUMMARY:
In recent years, the trend is for the patient to participate in their care. The development of new technologies together with the opportunities to exchange information, control one's own health and the possibility of communication between the team and the patient have increased. This is a prospective study trying to know the real use of ICT (information and communication technologies) among our surgical patients, its ability to use it and the differences in terms of gender, age or social range between others

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years scheduled to surgery in our Department

Exclusion Criteria:

* Inability to read
* Inability to understand messages
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults in-hospital in our Department of Surgery patients, scheduled to any surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Use of ITC | 6-12 months
  Number of patients with access to Internet
Rate of Use Health applications | 6-12 months
  Number of patients with an Health app

SECONDARY OUTCOMES:
Level of acceptance of ITC | 6-12 months
  Degree of ITC use on a diary basis

CONTACTS AND LOCATIONS:
Overall Officials: Jose-M Ramirez, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Hospital Clinico Lozano Blesa, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindberg B, Nilsson C, Zotterman D, Soderberg S, Skar L. Using Information and Communication Technology in Home Care for Communication between Patients, Family Members, and Healthcare Professionals: A Systematic Review. Int J Telemed Appl. 2013;2013:461829. doi: 10.1155/2013/461829. Epub 2013 Apr 10. PMID 23690763
- [Background] Holthe T, Halvorsrud L, Karterud D, Hoel KA, Lund A. Usability and acceptability of technology for community-dwelling older adults with mild cognitive impairment and dementia: a systematic literature review. Clin Interv Aging. 2018 May 4;13:863-886. doi: 10.2147/CIA.S154717. eCollection 2018. PMID 29765211
- [Background] Montroni I, Ugolini G, Saur NM, Spinelli A, Rostoft S, Millan M, Wolthuis A, Daniels IR, Hompes R, Penna M, Furst A, Papamichael D, Desai AM, Cascinu S, Gerard JP, Myint AS, Lemmens VEPP, Berho M, Lawler M, De Liguori Carino N, Potenti F, Nanni O, Altini M, Beets G, Rutten H, Winchester D, Wexner SD, Audisio RA. Personalized management of elderly patients with rectal cancer: Expert recommendations of the European Society of Surgical Oncology, European Society of Coloproctology, International Society of Geriatric Oncology, and American College of Surgeons Commission on Cancer. Eur J Surg Oncol. 2018 Nov;44(11):1685-1702. doi: 10.1016/j.ejso.2018.08.003. Epub 2018 Aug 15. PMID 30150158
- [Background] Anderberg P, Skar L, Abrahamsson L, Berglund JS. Older People's Use and Nonuse of the Internet in Sweden. Int J Environ Res Public Health. 2020 Dec 4;17(23):9050. doi: 10.3390/ijerph17239050. PMID 33291654
- [Background] Tomas CC, Oliveira E, Sousa D, Uba-Chupel M, Furtado G, Rocha C, Teixeira A, Ferreira P, Alves C, Gisin S, Catarino E, Carvalho N, Coucelo T, Bonfim L, Silva C, Franco D, Gonzalez JA, Jardim HG, Silva R, Baixinho CL, Presado M feminineH, Marques M feminineF, Cardoso ME, Cunha M, Mendes J, Xavier A, Galhardo A, Couto M, Frade JG, Nunes C, Mesquita JR, Nascimento MS, Goncalves G, Castro C, Martires A, Monteiro M feminineJ, Rainho C, Caballero FP, Monago FM, Guerrero JT, Monago RM, Trigo AP, Gutierrez ML, Milanes GM, Reina MG, Villanueva AG, Pinero AS, Aliseda IR, Ramirez FB, Ribeiro A, Quelhas A, Manso C, Caballero FP, Guerrero JT, Monago FM, Santos RB, Jimenez NR, Nunez CG, Gomez IR, Fernandez M feminineJL, Marquez LA, Moreno AL, Huertas M feminineJT, Ramirez FB, Seabra D, Salvador M feminineC, Braga L, Parreira P, Salgueiro-Oliveira A, Arreguy-Sena C, Oliveira BF, Henriques M feminineA, Santos J, Lebre S, Marques A, Festas C, Rodrigues S, Ribeiro A, Lumini J, Figueiredo AG, Hernandez-Martinez FJ, Campi L, Quintana-Montesdeoca M feminineP, Jimenez-Diaz JF, Rodriguez-De-Vera BC, Parente A, Mata M feminineA, Pereira AM feminine, Fernandes A, Bras M, Pinto M feminineR, Parreira P, Basto ML, Rei AC, Monico LM, Sousa G, Morna C, Freitas O, Freitas G, Jardim A, Vasconcelos R, Horta LG, Rosa RS, Kranz LF, Nugem RC, Siqueira MS, Bordin R, Kniess R, Lacerda JT, Guedes J, Machado I, Almeida S, Zilhao A, Alves H, Ribeiro O, Amaral AP, Santos A, Monteiro J, Rocha M feminineC, Cruz R, Amaral AP, Lourenco M, Rocha M feminineC, Cruz R, Antunes S, Mendonca V, Andrade I, Osorio N, Valado A, Caseiro A, Gabriel A, Martins AC, Mendes F, Cabral L, Ferreira M, Goncalves A, Luz TD, Luz L, Martins R, Morgado A, Vale-Dias ML, Porta-Nova R, Fleig TC, Reuter EM, Froemming MB, Guerreiro SL, Carvalho LL, Guedelha D, Coelho P, Pereira A, Calha A, Cordeiro R, Goncalves A, Certo A, Galvao A, Mata M feminineA, Welter A, Pereira E, Ribeiro S, Kretzer M, Jimenez-Diaz JF, Jimenez-Rodriguez C, Hernandez-Martinez FJ, Rodriguez-De-Vera BDC, Marques-Rodrigues A, Coelho P, Bernardes T, Pereira A, Sousa P, Filho JG, Nazario N, Kretzer M, Amaral O, Garrido A, Veiga N, Nunes C, Pedro AR, Pereira C, Almeia A, Fernandes HM, Vasconcelos C, Sousa N, Reis VM, Monteiro MJ, Mendes R, Pinto IC, Pires T, Gama J, Preto V, Silva N, Magalhaes C, Martins M, Duarte M, Paul C, Martin I, Pinheiro AA, Xavier S, Azevedo J, Bento E, Marques C, Marques M, Macedo A, Pereira AT, Almeida JP, Almeida A, Alves J, Sousa N, Saavedra F, Mendes R, Maia AS, Oliveira MT, Sousa AR, Ferreira PP, Lopes LS, Santiago EC, Monteiro S, Jesus A, Colaco A, Carvalho A, Silva RP, Cruz A, Ferreira A, Marques C, Figueiredo JP, Paixao S, Ferreira A, Lopes C, Moreira F, Figueiredo JP, Ferreira A, Ribeiro D, Moreira F, Figueiredo JP, Paixao S, Fernandes T, Amado D, Leal J, Azevedo M, Ramalho S, Mangas C, Ribeiro J, Goncalves R, Nunes AF, Tuna AR, Martins CR, Forte HD, Costa C, Tenedorio JA, Santana P, Andrade JA, Pinto JL, Campofiorito C, Nunes S, Carmo A, Kaliniczenco A, Alves B, Mendes F, Jesus C, Fonseca F, Gehrke F, Albuquerque C, Batista R, Cunha M, Madureira A, Ribeiro O, Martins R, Madeira T, Peixoto-Placido C, Santos N, Santos O, Bergland A, Bye A, Lopes C, Alarcao V, Goulao B, Mendonca N, Nicola P, Clara JG, Gomes J, Querido A, Tomas C, Carvalho D, Cordeiro M, Rosa MC, Marques A, Brandao D, Ribeiro O, Araujo L, Paul C, Minghelli B, Richaud S, Mendes AL, Marta-Simoes J, Trindade IA, Ferreira C, Carvalho T, Cunha M, Pinto-Gouveia J, Fernandes MC, Rosa RS, Nugem RC, Kranz LF, Siqueira MS, Bordin R, Martins AC, Medeiros A, Pimentel R, Fernandes A, Mendonca C, Andrade I, Andrade S, Menezes RL, Bravo R, Miranda M, Ugartemendia L, Tena JM feminine, Perez-Caballero FL, Fuentes-Broto L, Rodriguez AB, Carmen B, Carneiro MA, Domingues JN, Paixao S, Figueiredo J, Nascimento VB, Jesus C, Mendes F, Gehrke F, Alves B, Azzalis L, Fonseca F, Martins AR, Nunes A, Jorge A, Veiga N, Amorim A, Silva A, Martinho L, Monteiro L, Silva R, Coelho C, Amaral O, Coelho I, Pereira C, Correia A, Rodrigues D, Marante N, Silva P, Carvalho S, Araujo AR, Ribeiro M, Coutinho P, Ventura S, Roque F, Calvo C, Reses M, Conde J, Ferreira A, Figueiredo J, Silva D, Seica L, Soares R, Mourao R, Kraus T, Abreu AC, Padilha JM, Alves JM, Sousa P, Oliveira M, Sousa J, Novais S, Mendes F, Pinto J, Cruz J, Marques A, Duarte H, Dixe MDA, Sousa P, Cruz I, Bastos F, Pereira F, Carvalho FL, Oliveira TT, Raposo VR, Rainho C, Ribeiro JC, Barroso I, Rodrigues V, Neves C, Oliveira TC, Oliveira B, Morais M feminineC, Baylina P, Rodrigues R, Azeredo Z, Vicente C, Dias H, Sim-Sim M, Parreira P, Salgueiro-Oliveira A, Castilho A, Melo R, Graveto J, Gomes J, Vaquinhas M, Carvalho C, Monico L, Brito N, Sarroeira C, Amendoeira J, Cunha F, Candido A, Fernandes P, Silva HR, Silva E, Barroso I, Lapa L, Antunes C, Goncalves A, Galvao A, Gomes M feminineJ, Escanciano SR, Freitas M, Parreira P, Maroco J, Fernandes AR, Cabral C, Alves S, Sousa P, Ferreira A, Principe F, Seppanen UM, Ferreira M, Carvalhais M, Silva M, Ferreira M, Silva J, Neves J, Costa D, Santos B, Duarte S, Marques S, Ramalho S, Mendes I, Louro C, Menino E, Dixe M, Dias SS, Cordeiro M, Tomas C, Querido A, Carvalho D, Gomes J, Valim FC, Costa JO, Bernardes LG, Prebianchi H, Rosa MC, Goncalves N, Martins MM, Kurcgant P, Vieira A, Bento S, Deodato S, Rabiais I, Reis L, Torres A, Soares S, Ferreira M, Graca P, Leitao C, Abreu R, Bellem F, Almeida A, Ribeiro-Varandas E, Tavares A, Frade JG, Henriques C, Menino E, Louro C, Jordao C, Neco S, Morais C, Ferreira P, Silva CR, Brito A, Silva A, Duarte H, Dixe MDA, Sousa P, Postolache G, Oliveira R, Moreira I, Pedro L, Vicente S, Domingos S, Postolache O, Silva D, Filho JG, Nazario N, Kretzer M, Schneider D, Marques FM, Parreira P, Carvalho C, Monico LM, Pinto C, Vicente S, Breda SJ, Gomes JH, Melo R, Parreira P, Salgueiro A, Graveto J, Vaquinhas M, Castilho A, Jesus A, Duarte N, Lopes JC, Nunes H, Cruz A, Salgueiro-Oliveira A, Parreira P, Basto ML, Braga LM, Ferreira A, Araujo B, Alves JM, Ferreira M, Carvalhais M, Silva M, Novais S, Sousa AS, Ferrito C, Ferreira PL, Rodrigues A, Ferreira M, Oliveira I, Ferreira M, Neves J, Costa D, Duarte S, Silva J, Santos B, Martins C, Macedo AP, Araujo O, Augusto C, Braga F, Gomes L, Silva MA, Rosario R, Pimenta L, Carreira D, Teles P, Barros T, Tomas C, Querido A, Carvalho D, Gomes J, Cordeiro M, Carvalho D, Querido A, Tomas C, Gomes J, Cordeiro M, Jacome C, Marques A, Capelas S, Hall A, Alves D, Lousada M, Loureiro M feminineH, Camarneiro A, Silva M, Mendes A, Pedreiro A, G.Silva A, Coelho ES, Melo F, Ribeiro F, Torres R, Costa R, Pinho T, Jacome C, Marques A, Cruz B, Seabra D, Carreiras D, Ventura M, Cruz X, Brooks D, Marques A, Pinto MR, Parreira P, Lima-Basto M, Neves M, Monico LM, Bizarro C, Cunha M, Galhardo A, Margarida C, Amorim AP, Silva E, Cruz S, Padilha JM, Valente J, Guerrero JT, Caballero FP, Santos RB, Gonzalez EP, Monago FM, Ugalde LU, Velez MM, Tena MJ, Guerrero JT, Bravo R, Perez-Caballero FL, Becerra IA, Agudelo M feminineE, Acedo G, Bajo R, Malheiro I, Gaspar F, Barros L, Furtado G, Uba-Chupel M, Marques M, Rama L, Braga M, Ferreira JP, Teixeira AM feminine, Cruz J, Barbosa T, Simoes A, Coelho L, Rodrigues A, Jimenez-Diaz JF, Martinez-Hernandez F, Rodriguez-De-Vera B, Ferreira P, Rodrigues A, Ramalho A, Petrica J, Mendes P, Serrano J, Santo I, Rosado A, Mendonca P, Freitas K, Ferreira D, Brito A, Fernandes R, Gomes S, Moreira F, Pinho C, Oliveira R, Oliveira AI, Mendonca P, Casimiro AP, Martins P, Silva I, Evangelista D, Leitao C, Velosa F, Carecho N, Coelho L, Menino E, Dixe A, Catarino H, Soares F, Gama E, Gordo C, Moreira E, Midoes C, Santos M, Machado S, Oliveira VP, Santos M, Querido A, Dixe A, Marques R, Charepe Z, Antunes A, Santos S, Rosa MC, Rosa MC, Marques SF, Minghelli B, CaroMinghelli E, Luis M feminineJ, Brandao T, Mendes P, Marinho D, Petrica J, Monteiro D, Paulo R, Serrano J, Santo I, Monteiro L, Ramalho F, Santos-Rocha R, Morgado S, Bento T, Sousa G, Freitas O, Silva I, Freitas G, Morna C, Vasconcelos R, Azevedo T, Soares S, Pisco J, Ferreira PP, Olszewer EO, Oliveira MT, Sousa AR, Maia AS, Oliveira ST, Santos E, Oliveira AI, Maia C, Moreira F, Santos J, Mendes MF, Oliveira RF, Pinho C, Barreira E, Pereira A, Vaz JA, Novo A, Silva LD, Maia B, Ferreira E, Pires F, Andrade R, Camarinha L, Silva LD, Maia B, Ferreira E, Pires F, Andrade R, Camarinha L, Cesar AF, Poco M, Ventura D, Loura R, Gomes P, Gomes C, Silva C, Melo E, Lindo J, Domingos J, Mendes Z, Poeta S, Carvalho T, Tomas C, Catarino H, Dixe M feminineA, Ramalho A, Rosado A, Mendes P, Paulo R, Garcia I, Petrica J, Rodrigues S, Meneses R, Afonso C, Faria L, Seixas A, Cordeiro M, Granjo P, Gomes JC, Souza NR, Furtado GE, Rocha SV, Silva P, Carvalho J, Morais MA, Santos S, Lebre P, Antunes A, Calha A, Xavier A, Cunha M, Pinto-Gouveia J, Alencar L, Cunha M, Madureira A, Cardoso I, Galhardo A, Daniel F, Rodrigues V, Luz L, Luz T, Ramos MR, Medeiros DC, Carmo BM, Seabra A, Padez C, Silva MC, Rodrigues A, Coelho P, Coelho A, Caminha M, Matheus F, Mendes E, Correia J, Kretzer M, Hernandez-Martinez FJ, Jimenez-Diaz JF, Rodriguez-De-Vera BC, Jimenez-Rodriguez C, Armas-Gonzalez Y, Rodrigues C, Pedroso R, Apolinario-Hagen J, Vehreschild V, Veloso M, Magalhaes C, Cabral I, Ferraz M, Nave F, Costa E, Matos F, Pacheco J, Dias A, Pereira C, Duarte J, Cunha M, Silva D, Monico LM, Alferes VR, Breda M feminineSJ, Carvalho C, Parreira PM, Morais M feminineC, Ferreira P, Pimenta R, Boavida J, Pinto IC, Pires T, Silva C, Ribeiro M, Viega-Branco M, Pereira F, Pereira AM feminine, Almeida FM, Estevez GL, Ribeiro S, Kretzer MR, Joao PV, Nogueira P, Novais S, Pereira A, Carneiro L, Mota M, Cruz R, Santiago L, Fontes-Ribeiro C, Furtado G, Rocha SV, Coutinho AP, Neto JS, Vasconcelos LR, Souza NR, Dantas E, Dinis A, Carvalho S, Castilho P, Pinto-Gouveia J, Sarreira-Santos A, Figueiredo A, Medeiros-Garcia L, Seabra P, Rodrigues R, Morais M feminineC, Fernandes PO, Santiago C, Figueiredo M feminineH, Basto ML, Guimaraes T, Coelho A, Graca A, Silva AM, Fonseca AR, Vale-Dias L, Minas B, Franco-Borges G, Simoes C, Santos S, Serra A, Matos M, Jesus L, Tavares AS, Almeida A, Leitao C, Varandas E, Abreu R, Bellem F, Trindade IA, Ferreira C, Pinto-Gouveia J, Marta-Simoes J, Amaral O, Miranda C, Guimaraes P, Goncalves R, Veiga N, Pereira C, Fleig TC, San-Martin EA, Goulart CL, Schneiders PB, Miranda NF, Carvalho LL, Silva AG, Topa J, Nogueira C, Neves S, Ventura R, Nazare C, Brandao D, Freitas A, Ribeiro O, Paul C, Merce C, Branco M, Almeida P, Nascimento D, Pereira J, Catela D, Rafael H, Reis AC, Mendes A, Valente AR, Lousada M, Sousa D, Baltazar AL, Loureiro M feminineH, Oliveira A, Aparicio J, Marques A, Marques A, Oliveira A, Neves J, Ayoub R, Sousa L, Marques-Vieira C, Severino S, Jose H, Cadorio I, Lousada M, Cunha M, Andrade D, Galhardo A, Couto M, Mendes F, Domingues C, Schukg S, Abrantes AM, Goncalves AC, Sales T, Teixo R, Silva R, Estrela J, Laranjo M, Casalta-Lopes J, Rocha C, Simoes PC, Sarmento-Ribeiro AB, Botelho M feminineF, Rosa MS, Fonseca V, Colaco D, Neves V, Jesus C, Hesse C, Rocha C, Osorio N, Valado A, Caseiro A, Gabriel A, Svensson L, Mendes F, Siba WA, Pereira C, Tomaz J, Carvalho T, Pinto-Gouveia J, Cunha M, Duarte D, Lopes NV, Fonseca-Pinto R, Duarte D, Lopes NV, Fonseca-Pinto R, Martins AC, Brandao P, Martins L, Cardoso M, Morais N, Cruz J, Alves N, Faria P, Mateus A, Morouco P, Alves N, Ferreira N, Mateus A, Faria P, Morouco P, Malheiro I, Gaspar F, Barros L, Parreira P, Cardoso A, Monico L, Carvalho C, Lopes A, Salgueiro-Oliveira A, Seixas A, Soares V, Dias T, Vardasca R, Gabriel J, Rodrigues S, Paredes H, Reis A, Marinho S, Filipe V, Lains J, Barroso J, Da Motta C, Carvalho CB, Pinto-Gouveia J, Peixoto E, Gomes AA, Costa V, Couto D, Marques DR, Leitao JA, Tavares J, Azevedo MH, Silva CF, Freitas J, Parreira P, Maroco J, Garcia-Gordillo MA, Collado-Mateo D, Chen G, Iezzi A, Sala JA, Parraca JA, Gusi N, Sousa J, Marques M, Jardim J, Pereira A, Simoes S, Cunha M, Sardo P, Guedes J, Lindo J, Machado P, Melo E, Carvalho CB, Benevides J, Sousa M, Cabral J, Da Motta C, Pereira AT, Xavier S, Azevedo J, Bento E, Marques C, Carvalho R, Marques M, Macedo A, Silva AM, Alves J, Gomes AA, Marques DR, Azevedo M feminineH, Silva C, Mendes A, Lee HD, Spolaor N, Oliva JT, Chung WF, Fonseca-Pinto R, Bairros K, Silva CD, Souza CA, Schroeder SS, Araujo E, Monteiro H, Costa R, Dias SS, Torgal J, Henriques CG, Santos L, Caceiro EF, Ramalho SA, Oliveira R, Afreixo V, Santos J, Mota P, Cruz A, Pimentel F, Marques R, Dixe M feminineA, Querido A, Sousa P, Benevides J, Da Motta C, Sousa M, Caldeira SN, Carvalho CB, Querido A, Tomas C, Carvalho D, Gomes J, Cordeiro M, Costa JO, Valim FC, Ribeiro LC, Charepe Z, Querido A, Figueiredo M feminineH, Aquino PS, Ribeiro SG, Pinheiro AB, Lessa PA, Oliveira MF, Brito LS, Pinto IN, Furtado AS, Castro RB, Aquino CQ, Martins ES, Pinheiro AB, Aquino PS, Oliveira LL, Pinheiro PC, Sousa CR, Freitas VA, Silva TM, Lima AS, Aquino CQ, Andrade KV, Oliveira CA, Vidal EF, Ganho-Avila A, Moura-Ramos M, Goncalves O, Almeida J, Silva A, Brito I, Amado J, Rodrigo A, Santos S, Gomes F, Rosa MC, Marques SF, Luis S, Cavalheiro L, Ferreira P, Goncalves R, Lopes RS, Cavalheiro L, Ferreira P, Goncalves R, Fiorin BH, Santos MS, Oliveira ES, Moreira RL, Oliveira EA, Filho BL, Palmeira L, Garcia T, Pinto-Gouveia J, Cunha M, Cardoso S, Palmeira L, Cunha M, Pinto-Gouveia J, Marta-Simoes J, Mendes AL, Trindade IA, Oliveira S, Ferreira C, Mendes AL, Marta-Simoes J, Trindade IA, Ferreira C, Nave F, Campos M, Gaudencio I, Martins F, Ferreira L, Lopes N, Fonseca-Pinto R, Rodrigues R, Azeredo Z, Vicente C, Silva J, Sousa P, Marques R, Mendes I, Rodrigues R, Azeredo Z, Vicente C, Vardasca R, Marques AR, Seixas A, Carvalho R, Gabriel J, Ferreira PP, Oliveira MT, Sousa AR, Maia AS, Oliveira ST, Costa PO, Silva MM, Arreguy-Sena C, Alvarenga-Martins N, Pinto PF, Oliveira DC, Parreira PD, Gomes AT, Braga LM, Araujo O, Lage I, Cabrita J, Teixeira L, Marques R, Dixe M feminineA, Querido A, Sousa P, Silva S, Cordeiro E, Pimentel J, Ferro-Lebres V, Souza JA, Tavares M, Dixe M feminineA, Sousa P, Passadouro R, Peralta T, Ferreira C, Lourenco G, Serrano J, Petrica J, Paulo R, Honorio S, Mendes P, Simoes A, Carvalho L, Pereira A, Silva S, Sousa P, Padilha JM, Figueiredo D, Valente C, Marques A, Ribas P, Sousa J, Brandao F, Sousa C, Martins M, Sousa P, Marques R, Mendes F, Fernandes R, Martins E, Magalhaes C, Araujo P, Grande C, Mata M feminineA, Vieitez JG, Bianchini B, Nazario N, Filho JG, Kretzer M, Costa T, Almeida A, Baffour G, Almeida A, Costa T, Baffour G, Azeredo Z, Laranjeira C, Guerra M, Barbeiro AP, Ferreira R, Lopes S, Nunes L, Mendes A, Martins J, Schneider D, Kretzer M, Magajewski F, Soares C, Marques A, Batista M, Castuera RJ, Mesquita H, Faustino A, Santos J, Honorio S, Vizzotto BP, Frigo L, Pivetta HF, Sardo D, Martins C, Abreu W, Figueiredo M feminineC, Batista M, Jimenez-Castuera R, Petrica J, Serrano J, Honorio S, Paulo R, Mendes P, Sousa P, Marques R, Faustino A, Silveira P, Serrano J, Paulo R, Mendes P, Honorio S, Oliveira C, Bastos F, Cruz I, Rodriguez CK, Kretzer MR, Nazario NO, Cruz P, Vaz DC, Ruben RB, Avelelas F, Silva S, Campos M feminineJ, Almeida M, Goncalves L, Antunes L, Sardo P, Guedes J, Simoes J, Machado P, Melo E, Cardoso S, Santos O, Nunes C, Loureiro I, Santos F, Alves G, Soar C, Marsi TO, Silva E, Pedrosa D, Leca A, Silva D, Galvao A, Gomes M, Fernandes P, None A, Combadao J, Ramalhete C, Figueiredo P, Caeiro P, Fontana KC, Lacerda JT, Machado PO, Borges R, Barbosa F, Sa D, Brunhoso G, Aparicio G, Carvalho A, Garcia AP, Fernandes PO, Santos A, Veiga N, Bras C, Carvalho I, Batalha J, Gloria M, Bexiga F, Coelho I, Amaral O, Pereira C, Pinho C, Paraiso N, Oliveira AI, Lima CF, Dias AP, Silva P, Espada M, Marques M, Pereira A, Pereira AM feminine, Veiga-Branco M feminine, Pereira F, Ribeiro M, Lima V, Oliveira AI, Pinho C, Cruz G, Oliveira RF, Barreiros L, Moreira F, Camarneiro A, Loureiro M feminineH, Silva M, Duarte C, Jesus A, Cruz A, Mota M, Novais S, Nogueira P, Pereira A, Carneiro L, Joao PV, Lima TM, Salgueiro-Oliveira A, Vaquinhas M, Parreira P, Melo R, Graveto J, Castilho A, Gomes JH, Medina MS, Blanco VG, Santos O, Lopes E, Virgolino A, Dinis A, Ambrosio S, Almeida I, Marques T, Heitor M feminineJ, Garcia-Gordillo MA, Collado-Mateo D, Olivares PR, Parraca JA, Sala JA, Castilho A, Graveto J, Parreira P, Oliveira A, Gomes JH, Melo R, Vaquinhas M, Cheio M, Cruz A, Pereira OR, Pinto S, Oliveira A, Manso MC, Sousa C, Vinha AF, Machado M feminineM, Vieira M, Fernandes B, Tomas T, Quirino D, Desouzart G, Matos R, Bordini M, Mouroco P, Matos AR, Serapioni M, Guimaraes T, Fonseca V, Costa A, Ribeiro J, Lobato J, Martin IZ, Bjorklund A, Tavares AI, Ferreira P, Passadouro R, Morgado S, Tavares N, Valente J, Martins AC, Araujo P, Fernandes R, Mendes F, Magalhaes C, Martins E, Mendes P, Paulo R, Faustino A, Mesquita H, Honorio S, Batista M, Lacerda JT, Ortiga AB, Calvo M feminineC, Natal S, Pereira M, Ferreira M, Prata AR, Nelas P, Duarte J, Carneiro J, Oliveira AI, Pinho C, Couto C, Oliveira RF, Moreira F, Maia AS, Oliveira MT, Sousa AR, Ferreira PP, Souza GM, Almada LF, Conceicao MA, Santiago EC, Rodrigues S, Domingues G, Ferreira I, Faria L, Seixas A, Costa AR, Jesus A, Cardoso A, Meireles A, Colaco A, Cruz A, Vieira VL, Vincha KR, Cervato-Mancuso AM feminine, Faria M, Reis C, Cova MP, Ascenso RT, Almeida HA, Oliveira EG, Santana M, Pereira R, Oliveira EG, Almeida HA, Ascenso RT, Jesus R, Tapadas R, Tim-Tim C, Cezanne C, Lagoa M, Dias SS, Torgal J, Lopes J, Almeida H, Amado S, Carrao L, Cunha M, Saboga-Nunes L, Albuquerque C, Ribeiro O, Oliveira S, Morais M feminineC, Martins E, Mendes F, Fernandes R, Magalhaes C, Araujo P, Pedro AR, Amaral O, Escoval A, Assuncao V, Luis H, Luis L, Apolinario-Hagen J, Vehreschild V, Fotschl U, Lirk G, Martins AC, Andrade I, Mendes F, Mendonca V, Antunes S, Andrade I, Osorio N, Valado A, Caseiro A, Gabriel A, Martins AC, Mendes F, Silva PA, Monico LM, Parreira PM, Carvalho C, Carvalho C, Parreira PM, Monico LM, Ruivo J, Silva V, Sousa P, Padilha JM, Ferraz V, Aparicio G, Duarte J, Vasconcelos C, Almeida A, Neves J, Correia T, Amorim H, Mendes R, Saboga-Nunes L, Cunha M, Albuquerque C, Pereira ES, Santos LS, Reis AS, Silva HR, Rombo J, Fernandes JC, Fernandes P, Ribeiro J, Mangas C, Freire A, Silva S, Francisco I, Oliveira A, Catarino H, Dixe M feminineA, Louro M feminineC, Lopes S, Dixe A, Dixe M feminineA, Menino E, Catarino H, Soares F, Oliveira AP, Gordo S, Kraus T, Tomas C, Queiros P, Rodrigues T, Sousa P, Frade JG, Lobao C, Moura CB, Dreyer LC, Meneghetti V, Cabral PP, Pinto F, Sousa P, Esteves M feminineR, Galvao S, Tytgat I, Andrade I, Osorio N, Valado A, Caseiro A, Gabriel A, Martins AC, Mendes F, Casas-Novas M, Bernardo H, Andrade I, Sousa G, Sousa AP, Rocha C, Belo P, Osorio N, Valado A, Caseiro A, Gabriel A, Martins AC, Mendes F, Martins F, Pulido-Fuentes M, Barroso I, Cabral G, Monteiro MJ, Rainho C, Prado A, Carvalho YM, Campos M, Moreira L, Ferreira J, Teixeira A, Rama L, Campos M, Moreira L, Ferreira J, Teixeira A, Rama L. Proceedings of the 3rd IPLeiria's International Health Congress : Leiria, Portugal. 6-7 May 2016. BMC Health Serv Res. 2016 Jul 6;16 Suppl 3(Suppl 3):200. doi: 10.1186/s12913-016-1423-5. PMID 27409075
- [Background] de Veer AJ, Peeters JM, Brabers AE, Schellevis FG, Rademakers JJ, Francke AL. Determinants of the intention to use e-Health by community dwelling older people. BMC Health Serv Res. 2015 Mar 15;15:103. doi: 10.1186/s12913-015-0765-8. PMID 25889884
- [Background] Ball C, Francis J, Huang KT, Kadylak T, Cotten SR, Rikard RV. The Physical-Digital Divide: Exploring the Social Gap Between Digital Natives and Physical Natives. J Appl Gerontol. 2019 Aug;38(8):1167-1184. doi: 10.1177/0733464817732518. Epub 2017 Sep 19. PMID 29165009